CLINICAL TRIAL: NCT04148430
Title: A Phase II Study of IL-1 Receptor Antagonist Anakinra to Prevent Severe Neurotoxicity and Cytokine Release Syndrome in Patients Receiving CD19-Specific Chimeric Antigen Receptor (CAR) T Cells
Brief Title: A Study of Anakinra to Prevent or Treat Severe Side Effects for Patients Receiving CAR-T Cell Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-168
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: B Cell ALL; B-Cell Lymphoma; B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (CART Cell Group) (Experimental): Cohort 1 Patients will receive anakinra 100mg s.c. every 12 hours starting on day 2 post CAR T cell infusion, or after 2 documented fevers of ≥38.5° C prior to day 2, whichever time point is earlier. Anakinra will be continued for 10 days.
  Cohort 2 Patients will receive anakinra 100mg s.c. daily on day 0 of T cell infusion, and continue anakinra daily for 7 days
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — 100mg subcutaneous

SUMMARY:
This study is being done to see if the investigational drug, anakinra, prevent or reverse the severe side effects caused by CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age >/= 18) with a diagnosis of relapsed CD19+ B-cell ALL, MCL, or NHL receiving commercially approved CD19-specific CAR T cells (e.g. tisagenleuleucel, axicabtagene, brexucabtagene autoleucel, etc) are eligible for the study

Exclusion Criteria:

* Patients with uncontrolled systemic fungal and bacterial infections
* Patients with known hypersensitivity to E. coli-derived proteins
* Women of childbearing potential must have a negative serum or urine pregnancy test (women who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Arm 1 (CAR T Cell Group) Rate of Severe Neurotoxicities | 4 weeks
  Determine the rate of severe neurotoxicities, >/= Grade 3 or any grade seizure, within the first 4 weeks of treatment with prophylactic use of anakinra in participants receiving CD19-specific CAR T cells
Arm 2 (COVID-19 Group) proportion of patients able to avoid death or mechanical ventilation | 28 days from the start of treatment
  proportion of patients able to avoid death or mechanical ventilation within 28 days from the start of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Hackensack Meridian Health (Data collection only), Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Danish H, Santomasso BD. Neurotoxicity Biology and Management. Cancer J. 2021 Mar-Apr 01;27(2):126-133. doi: 10.1097/PPO.0000000000000507. PMID 33750072
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org